CLINICAL TRIAL: NCT06727201
Title: The Effect of Ondansetron on the Total Consumption of Norepinephrine Infusion Used to Prevent Spinal Anaesthesia Induced Hypotention in Cesarean Section.
Brief Title: Role of Ondansetron in Spinal Anaesthesia Induced Hypotension
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Waleed Tarek Farouk, Resident, Assiut University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Role of ondansetron
Record Dates: First submitted 2024-11-28; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Spinal Anaesthesia Induced Hypotension
Keywords: Ondansetron; Spinal anaethesia; Hypotension; Norepinephrine
MeSH Terms: conditions — Hypotension | interventions — Ondansetron; Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ondansetron (Zofran) (Active Comparator): Ondansetron will be given intravenously in a dose of 0.1mg/kg 10 minutes before spinal anaesthesia as single shot
  Interventions: Drug: Ondansetron (Zofran)
- Saline placebo (Placebo Comparator): Normal saline will be administered by intravenous infusion 10 minutes before spinal anaesthesia
  Interventions: Drug: Saline (NaCl 0,9 %) (placebo)

INTERVENTIONS:
Drug: Ondansetron (Zofran) — Ondansetron will be given intravenously in a dose of 0.1mg/kg 10 minutes before spinal anaesthesia as single shot.
  Arms: Ondansetron (Zofran)
Drug: Saline (NaCl 0,9 %) (placebo) — normal saline infusion will be given intravenously 10 minutes before spinal anaesthesia
  Arms: Saline placebo

SUMMARY:
The objective of this study is to determine the effect of ondansetron on the total consumption of norepinephrine infusion needed to prevent spinal anaesthesia induced hypotension in cesarean section.

DETAILED DESCRIPTION:
Ondansetron has been reported to attenuate the incidence of spinal anaesthesia-induced hypotension (SAIH) and norepinephrine requirement during caesarean section.

The mechanism of hypotension following spinal anaesthesia involves the reduction in vascular resistance caused by the sympathetic block and the activation of the Bezold-Jarisch reflex, leading to vasodilation and hypotension. Peripheral serotonin receptors, 5-Hydroxytryptamine3 (5HT3), are required for the activation of the Bezold-Jarisch reflex. In a rabbit model, a 5-HT3 receptor antagonist was reported to suppress bradycardia and hypotension by preventing the Bezold-Jarisch reflex.

ELIGIBILITY:
Inclusion Criteria:

* Age from 19 to 40 years old.
* Singleton pregnancies with a gestational age of at least 37 weeks.
* pregnant women are scheduled for elective caesarean delivery.
* Patients with stable vital signs.
* Patients with normal laboratory investigations.
* patients undergoing spinal anaesthesia for caesarean delivery via Pfannenstiel incision with exteriorizaion of the uterus.

Exclusion Criteria:

* Patient's refusal.
* Age < 19 or > 40 years.
* Height<150 cm, weight < 60 kg, body mass index (BMI) ≥40 kg/m2.
* Contraindications to spinal anaesthesia (Coagulopathy, increased intracranial pressure, or local skin infection).
* Patients with cardiac morbidities.
* hypertensive disorders of pregnancy as pre-eclampsia.
* peripartum bleeding.
* Patients with respiratory morbidities.
* Convulsions.
* Bleeding diathesis.
* Known allergy to any drugs used in this study.

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 160 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Total consumption of norepinephrine during the whole surgical procedure. | Just after subarachnoid block till the end of surgery
  Comparison between total amount of vassopressor used to maintain normal blood pressure in both groups of study

SECONDARY OUTCOMES:
Incidence of hypotension, hemodynamic data and postoperative complications(nausea,vomiting,hypertension and bradycardia). | Just after subarachnoid block till 24 hours postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed H Bakri, professor, Study Director — Assiut University; Ola M Wahba, A.professor, Study Director — Assiut University; Abdelrahman H Mohammed, A.professor, Study Director — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt

REFERENCES:
- [Result] Sheng ZM, Sun HQ, Mao JQ, Liu J, Liang G, Mei Z. Comparative dose-response study on the infusion of norepinephrine combined with intravenous ondansetron versus placebo for preventing hypotension during spinal anesthesia for cesarean section: a randomised controlled trial. Int J Surg. 2024 Feb 1;110(2):832-838. doi: 10.1097/JS9.0000000000000920. PMID 38000073